CLINICAL TRIAL: NCT07184593
Title: Validation of a Point-of-care Device for Rapid Bedside Measurement of Circulating Nucleosome Levels in Critically Ill Patients and Study of Its Relevance to Prognostication
Brief Title: Nucleosome Monitoring Relevance for Outcome Prediction in Critically Ill Patients
Acronym: NuROPI
Status: Not yet recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Charles Dehout, Attending physician, PhD student, Erasme University Hospital
Other Study IDs: HUB2025237
Record Dates: First submitted 2025-08-26; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sepsis; Septic Shock; Cardiac Arrest (CA); Pancreatitis; Acute Brain Injury; Trauma Blunt; Cardiogenic Shock
Keywords: nucleosome; septic shock; Histones; Cardiac Arrest; Cardiogenic shock; Trauma; Acute brain injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Heart Arrest; Pancreatitis; Brain Injuries; Wounds, Nonpenetrating; Shock, Cardiogenic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and cerebrospinal fluid of patients at 5 different timepoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Sepsis: As defined by sepsis-3 definition (excluding septic shock, around 30 patients)
- Septic shock: as defined per SEPSIS-3 definition (around 30 patients)
- Cardiogenic shock: classified as at least SCAI stage C (approximately 10 patients)
- Severe trauma: Requiring at least 4 units of red blood cells within 6 hours post-admission (approximately 10 patients)
- Acute brain injury: requiring invasive neuromonitoring (approximately 20 patients)
- Post-cardiac arrest: With at least 15 minutes of no or low perfusion (intra or extra hospital setting) (approximately 20 patients)
- Severe acute pancreatitis: requiring ICU management (approximately 10 patients)

SUMMARY:
The goal of this observational study is to evaluate whether whole blood H3.1 nucleosome levels can predict 30-day mortality in adult critically ill patients admitted to the ICU with conditions such as sepsis, septic shock, cardiogenic shock, severe trauma, post-cardiac arrest, acute brain injury, or severe acute pancreatitis.

The main questions it aims to answer are:

Do initial whole blood H3.1 nucleosome levels predict 30-day mortality in critically ill patients?

Are whole blood nucleosome measurements using a novel point-of-care device correlated with traditional plasma chemiluminescence immunoassays (ChLIA)?

If there is a comparison group: Researchers will compare point-of-care whole blood nucleosome results with plasma ChLIA assays to see if the device provides reliable and feasible bedside measurements.

Participants will:

Provide blood samples at admission, 6h, Day 1, Day 3, and Day 7 for nucleosome analysis.

Undergo point-of-care H3.1 nucleosome measurement and parallel plasma storage for ChLIA testing.

(If applicable, in acute brain injury patients with external ventricular drains) provide daily cerebrospinal fluid samples until Day 5, only if otherwise discarded.

Have standard ICU data (SOFA, SAPS II, etc.) collected as part of routine care.

DETAILED DESCRIPTION:
The NuROPI study is a prospective, observational, non-interventional, monocentric study conducted in the Intensive Care Unit (ICU) of Erasme Hospital, Brussels. It aims to evaluate the association between initial levels of H3.1 nucleosomes in whole blood and 30-day mortality in critically ill patients, and to validate a novel point-of-care device for nucleosome measurement against standard chemiluminescence immunoassay (ChLIA) performed on plasma.

Inclusion requires the presence of an arterial or central venous catheter for blood sampling. Exclusion criteria include age <18, life expectancy <24 hours, therapeutic limitations, active cancer, absence of vascular access, ICU stay >24h before screening, or prior inclusion. Blood will be sampled at five predefined timepoints: admission (H0), 6 hours (H6), Day 1 (D1), Day 3 (D3), and Day 7 (D7). At each timepoint, four 5 mL blood tubes will be collected during routine care, and a 20 µL aliquot will be used for immediate point-of-care H3.1 measurement. Plasma will be extracted and stored for delayed ChLIA analysis. In patients with acute brain injury and an external ventricular drain (EVD), cerebrospinal fluid (CSF) will be sampled daily until Day 5, but only if the fluid is otherwise intended to be discarded. The study seeks to establish whether nucleosome levels can serve as a biomarker for prognosis and patient stratification in critical illness.

Standard ICU data such as SOFA scores and SAPS II will be recorded, as is already routinely done in some registries like Epimed.

Data will be entered into RedCap by the research team and the investigators.

The study population will consist of 130 adult critically ill patients admitted to the Intensive Care Unit (ICU) of Erasme Hospital. Eligible participants must be 18 years or older and admitted to the ICU within the past 24 hours. All patients must have arterial or central venous access for blood sampling. The population will include a diverse group of critically ill individuals representing various acute conditions commonly encountered in intensive care:

* Sepsis, as defined by SEPSIS-3 criteria (approximately 30 patients)
* Septic shock, per SEPSIS-3 (approximately 30 patients)
* Cardiogenic shock, classified as at least SCAI stage C (approximately 10 patients)
* Severe trauma, requiring at least 4 units of red blood cells within 6 hours post-admission (approximately 10 patients)
* Acute brain injury, requiring invasive neuromonitoring (approximately 20 patients)
* Post-cardiac arrest, with at least 15 minutes of no or low perfusion (approximately 20 patients)
* Severe acute pancreatitis, requiring ICU management (approximately 10 patients) This heterogeneous ICU population is specifically chosen to evaluate the relevance of H3.1 nucleosome levels across multiple critical illness etiologies.

Objectives

Primary

- To evaluate the association between initial levels of H3.1 nucleosomes in whole blood and 30-day mortality in a cohort of critically ill patients.

Secondary

* To assess the correlation between nucleosome levels measured in whole blood at the point of care and traditional chemiluminescence immunoassays performed on plasma.
* To validate the feasibility and reliability of a novel point-of-care device for rapid nucleosome quantification.
* To determine whether nucleosome measurement is relevant across a variety of critical conditions (e.g., sepsis, septic shock, cardiogenic shock, severe trauma, cardiac arrest, acute brain injury, severe acute pancreatitis)

ELIGIBILITY:
Inclusion Criteria:

* Admission to the intensive care unit (ICU) within the past 24 hours.
* Patient must meet one of the following conditions:

Sepsis, defined according to SEPSIS-3 criteria.

Septic shock, defined according to SEPSIS-3 criteria.

Cardiogenic shock, classified as Stage C according to the Society for Cardiovascular Angiography and Interventions (SCAI).

Severe trauma requiring transfusion of four or more units of red blood cells within six hours.

Acute brain injury requiring invasive neuromonitoring.

Post-cardiac arrest with at least 15 minutes of no or low perfusion.

Severe acute pancreatitis requiring ICU-level care.

- Presence of an arterial or central venous catheter to allow blood sampling.

Exclusion Criteria

* Patient who has expressed opposition to participate.
* Age younger than 18 years.
* Imminent death with an expected survival of less than 24 hours.
* Presence of therapeutic limitations (e.g., no indication for intubation).
* Active cancer.
* Absence of the required vascular access.
* ICU admission longer than 24 hours prior to screening.
* Readmission of a previously enrolled patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 130 adult critically ill patients admitted to the Intensive Care Unit (ICU) of Erasme Hospital. Eligible participants must be 18 years or older and admitted to the ICU within the past 24 hours. All patients must have arterial or central venous access for blood sampling. The population will include a diverse group of critically ill individuals representing various acute conditions commonly encountered in intensive care:
  Sepsis Septic shock Cardiogenic shock Severe trauma Acute brain injury Severe trauma Post-cardiac arrest shock Severe pancreatitis
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality D30 | 30 days
  To evaluate the association between initial levels of H3.1 nucleosomes in whole blood and 30-day mortality in a cohort of critically ill patients.

SECONDARY OUTCOMES:
Nucleosome measurement correlation between point-of-care and chemiluminescence immunoassays (ChLIA) | At each sampling time point - Day 0 (baseline), Hour 6, Day 1, Day 3, and Day 7
  To assess the correlation between nucleosome levels measured in whole blood at the point of care and traditional chemiluminescence immunoassays performed on plasma.
Cerebrospinal fluid (CSF) nucleosome levels | At each sampling time point - Day 0 (baseline), Hour 6, Day 1, Day 3, and Day 7
  Cerebrospinal fluid (CSF) nucleosome levels (in patients with invasive neuromonitoring), to explore their potential role as biomarkers in acute brain injury.
Prolonged organ failure | Up to 28 days after enrollment
  Defined as the need for organ support (e.g., mechanical ventilation, vasopressors, renal replacement therapy) persisting ≥7 consecutive days.
In-hospital mortality | Through hospital discharge (average of 14 days)
  All-cause mortality occurring during index hospitalization.

OTHER OUTCOMES:
Progression to chronic kidney disease (CKD) | At 3, 6, and 12 months after hospital discharge
  Defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m² persisting for ≥3 months, or requirement for chronic dialysis.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Su F, Moreau A, Savi M, Salvagno M, Annoni F, Zhao L, Xie K, Vincent JL, Taccone FS. Circulating Nucleosomes as a Novel Biomarker for Sepsis: A Scoping Review. Biomedicines. 2024 Jun 21;12(7):1385. doi: 10.3390/biomedicines12071385. PMID 39061959
- [Background] Garcia B, Su F, Dewachter L, Wang Y, Li N, Remmelink M, Eycken MV, Khaldi A, Favory R, Herpain A, Moreau A, Moiroux-Sahraoui A, Manicone F, Annoni F, Shi L, Vincent JL, Creteur J, Taccone FS. Neutralization of extracellular histones by sodium-Beta-O-methyl cellobioside sulfate in septic shock. Crit Care. 2023 Nov 24;27(1):458. doi: 10.1186/s13054-023-04741-x. PMID 38001494
- [Background] Allam R, Kumar SV, Darisipudi MN, Anders HJ. Extracellular histones in tissue injury and inflammation. J Mol Med (Berl). 2014 May;92(5):465-72. doi: 10.1007/s00109-014-1148-z. Epub 2014 Apr 6. PMID 24706102
- [Background] Cheng Z, Abrams ST, Alhamdi Y, Toh J, Yu W, Wang G, Toh CH. Circulating Histones Are Major Mediators of Multiple Organ Dysfunction Syndrome in Acute Critical Illnesses. Crit Care Med. 2019 Aug;47(8):e677-e684. doi: 10.1097/CCM.0000000000003839. PMID 31162199
- [Background] Silk E, Zhao H, Weng H, Ma D. The role of extracellular histone in organ injury. Cell Death Dis. 2017 May 25;8(5):e2812. doi: 10.1038/cddis.2017.52. PMID 28542146
- [Background] Yang T, Peng J, Zhang Z, Chen Y, Liu Z, Jiang L, Jin L, Han M, Su B, Li Y. Emerging therapeutic strategies targeting extracellular histones for critical and inflammatory diseases: an updated narrative review. Front Immunol. 2024 Aug 14;15:1438984. doi: 10.3389/fimmu.2024.1438984. eCollection 2024. PMID 39206200
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185
- [Background] Ranieri VM, Thompson BT, Barie PS, Dhainaut JF, Douglas IS, Finfer S, Gardlund B, Marshall JC, Rhodes A, Artigas A, Payen D, Tenhunen J, Al-Khalidi HR, Thompson V, Janes J, Macias WL, Vangerow B, Williams MD; PROWESS-SHOCK Study Group. Drotrecogin alfa (activated) in adults with septic shock. N Engl J Med. 2012 May 31;366(22):2055-64. doi: 10.1056/NEJMoa1202290. Epub 2012 May 22. PMID 22616830
- [Background] Tindal EW, Armstead BE, Monaghan SF, Heffernan DS, Ayala A. Emerging therapeutic targets for sepsis. Expert Opin Ther Targets. 2021 Mar;25(3):175-189. doi: 10.1080/14728222.2021.1897107. Epub 2021 Apr 12. PMID 33641552
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338